CLINICAL TRIAL: NCT01628653
Title: Feasibility and Efficacy of the Ubiquitous Spaced Retrieval-based Memory Advancement and Rehabilitation Training (U-SMART) on Mild Cognitive Impairment
Brief Title: Ubiquitous Spaced Retrieval-based Memory Advancement and Rehabilitation Training
Acronym: U-SMART
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: KT Corporation (Industry)
Responsible Party: Principal Investigator, Ki Woong Kim, Professor, department of neuropsychiatry, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-2011-084
Record Dates: First submitted 2012-06-23; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild cognitive impairment; Cognitive rehabilitation; Cognitive therapy; Spaced retrieval Training; Alzheimer's disease; Memory enhancement; U-healthcare
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- U-SMART (Experimental): U-SMART (Ubiquitous Spaced Retrieval-based Memory Advancement and Rehabilitation Training)
  Interventions: Device: U-SMART

INTERVENTIONS:
Device: U-SMART — 4-weeks' training

SUMMARY:
The purpose of this study is to examine feasibility and efficacy of the Ubiquitous Spaced Retrieval-based Memory Advancement and Rehabilitation Training (U-SMART) in the elderly individuals with mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
The Spaced Retrieval-based Memory Advancement and Rehabilitation Training (SMART) which consisted of 24 one-hour face-to-face sessions (Lee, Park et al. 2009) was developed based on the spaced retrieval training (SRT), which was effective in improving memory retention span of very mild to mild Alzheimer's disease patients. The Ubiquitous SMART (U-SMART) by transforming the current SMART to a self-administered program using an application working on IPAD was developed, and was examined its feasibility and efficacy in the elderly individuals with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55-90
* Educational level above 1 year and confirmed literacy
* Diagnosed to mild cognitive impairment by International Working Group on Mild Cognitive Impairment
* Clinical Dementia Rating (CDR) of 0 or 0.5

Exclusion Criteria:

* Diagnosed to dementia by DSM-IV
* Evidence of delirium, confusion
* Any neurological conditions causing cognitive decline such as Parkinson's disease, brain hemorrhage, brain tumor, normal pressure hydrocephalus
* Evidence of severe cerebrovascular pathology
* History of loss-of-consciousness over 1 hour due to head trauma or repetitive head trauma of mild severity
* History of substance abuse or dependence such as alcohol
* Presence of depressive symptoms that could influence cognitive function
* Presence of medical comorbidities that could result in cognitive decline
* Use of medication that could influence cognitive function seriously

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
the five-point Likert scales for satisfaction and compliance | after 4-weeks treatment
  To evaluate the feasibility of the U-SMART, the five-point Likert scales for satisfaction and compliance were applied to all participants.
Word List Memory Test of the CERAD Neuropsychological Assessment Battery | after 4-weeks treatment
  To evaluate the efficacy of the U-SMART, the Word List Memory Test (WLMT) of the CERAD neuropsychological assessment battery was applied to all participants.

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | after 4-weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ki Woong Kim, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital, Seong-nam, Korea
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea